CLINICAL TRIAL: NCT00857285
Title: A Multi-center, Double Blind, Efficacy, and Safety Study of the Oral Angiotensin II Receptor Blocker "Olmesartan Medoxomil" Versus "Losartan" in Patients With Mild to Moderate Essential Hypertension
Brief Title: Olmesartan Medoxomil Versus Losartan in Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Taiwan Ltd. (Industry)
Responsible Party: Ammy Chou, Director, Daiichi Sankyo Taiwan Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSP-866/01
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2009-07-23 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Olmesartan Medoxomil; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): olmesartan medoxomil
  Interventions: Drug: olmesartan medoxomil
- 2 (Active Comparator): losartan potassium
  Interventions: Drug: losartan potassium

INTERVENTIONS:
Drug: olmesartan medoxomil — olmesartan medoxomil oral tablets, once daily for up to 12 weeks
  Arms: 1
Drug: losartan potassium — losartan oral tablets, once daily for up to 12 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to determine the efficacy and safety of oral administration of olmesartan medoxomil compared to losartan in subjects with mild to moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diastolic BP 95 mm Hg - 114 mm Hg inclusive
* No participation in any clinical trial for the last 3 months

Exclusion Criteria:

* Secondary hypertension
* Malignant hypertension
* Severe arterial hypertension
* Significant cardiovascular disease
* History or clinical evidence of cerebrovascular, gastrointestinal, hematological, hepatic disease, myocardial infarction, or severe liver disorder
* Clinical evidence of renal disease, poorly controlled diabetes, known malabsorption syndromes, psychiatric/emotional problems

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2002-05; Primary Completion 2003-08 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chung Shun Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 181 subjects were screened at 3 study sites in Taiwan from May 2002 to April 2003, and 51 subjects had dropped as screen failure.
Pre-assignment Details: After a taper off period for 1 week, if necessary, and a placebo run-in period for 2 weeks, 130 subjects were randomized to olmesartan 20mg and losartan 50mg by 1:1 ratio.
Groups:
- Losartan Potassium: losartan potassium oral tablets, once daily for up to 12 weeks
Period: Overall Study
Arm/Group | Olmesartan Medoxomil | Losartan Potassium
Started | 65 | 65
Completed | 53 | 59
Not Completed | 12 | 6
Not completed — Adverse Event | 4 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Randomization criteria not met | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olmesartan Medoxomil | Losartan Potassium | Total
Number analyzed (Participants) | 65 | 65 | 130
Age Continuous [Mean (Standard Deviation); unit: years] | 49.63 (10.69) | 48.34 (9.17) | 48.98 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 23 | 56
  Male | 32 | 42 | 74
Race/Ethnicity, Customized [Number; unit: participants]
  Taiwanese | 65 | 65 | 130
Region of Enrollment [Number; unit: participants]
  Taiwan | 65 | 65 | 130

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of Sitting dBP From Baseline to Week 12
Description: The difference in the sitting diastolic blood pressure (dBP) at trough, i.e. 24±2 hours after drug administration, from base line to Week 12.
Time Frame: Baseline to 12 weeks
Population: Four randomized subjects (3 in olmesartan, 1 in losartan) were excluded from the analysis due to a lack of post-treatment efficacy evaluation.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Olmesartan Medoxomil | Losartan Potassium
Number analyzed (Participants) | 62 | 64
mmHg | -14.80 (12.50) | -11.60 (9.46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No